CLINICAL TRIAL: NCT04385160
Title: Myeloproliferative Neoplasms (MPN) and COVID-19
Acronym: MPN-COVID
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: FROM - O-MPN-COVID-2020
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Myeloproliferative Neoplasm; COVID
Keywords: thrombosis
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An increased risk of both venous and arterial thromboembolism was noted in reports from SARS-CoV-2-infected patients in China and has been confirmed in autopsy findings from patients who experienced sudden death. Myeloproliferative Neoplasms (MPNs), which encompass polycythemia vera, essential thrombocythemia and primary myelofibrosis, are thrombophilic disorders with a natural propensity to thrombosis that is fuelled by the intrinsic activation of inflammatory cytokines. It therefore follows that an underlying diagnosis of MPN may increase the risk of worse clinical outcomes and death during periods of active Covid-19 disease. This ambispective, observational study aims to elucidate the key factors which affect the clinical course of patients with MPN who develop Covid-19 disease.

DETAILED DESCRIPTION:
This is an European multicenter observational study that will include around 550 MPN patients with a confirmed diagnosis of Covid-19 will be followed for at least one month. Detailed information on the clinical characteristics of these patients and their disease outcomes will be retrospectively and prospectively collected in a specific eCRF, including MPN characteristics, treatment and comorbidities pre-Covid-19, time of Covid-19 diagnosis, drugs/device used for the treatment of Covid-19, any change in MPN therapy, antithrombotic prophylaxis employed during the period of infection and - for hospitalised patients only - key blood and laboratory parameters. A particular focus will be on exploring final outcomes for patients in this study, most notably the incidence of fatal and non-fatal thrombotic events. Statistical analyses will also be performed looking for any independent factors that can significantly predict patient outcomes after Covid-19 diagnosis.

Ultimately, this project will provide important insights into disease severity and progression in patients with MPN and Covid-19 and uncover the key clinical factors which drive outcomes and mortality. Results may help clinicians better understand how patient characteristics and management decisions can impact on disease trajectory when MPN and Covid-19 collide.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed diagnosed of MPN according to WHO criteria
* Diagnosis of COVID-19 based by the positivity of oropharyngeal swab performed between 15 February 2020 up to 15 February 2022
* Signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myeloproliferative Neoplasm (Polycythemia Vera, Essential Polycythemia, Myelofibrosis) diagnosed with COVID-19 between 15 February 2020 and 15 February 2022
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
pulmonary embolism (PE) | 2 and a half months
  Incidence of cases of MPN patients with COVID-19 experiencing pulmonary embolism

SECONDARY OUTCOMES:
fatal or non fatal thrombotic event | 2 and a half months
  Incidence of cases reporting at least one fatal or non fatal thrombotic event reported in therapy of MPN, , with particular focus to those occurred during hospitalization
Continuous Positive Airway Pressure (CPAP) | 2 and a half months
  Incidence of cases reporting at least one COVID-19 worsening outcome as Continuous Positive Airway Pressure (CPAP)
invasive ventilation | 2 and a half months
  Incidence of cases reporting at least one COVID-19 worsening outcome as invasive ventilation
admission in Intensive Care Unit (ICU) | 2 and a half months
  Incidence of cases reporting at least one COVID-19 worsening outcome as Intensive Care Unit (ICU)
death | 2 and a half months
  incidence of death
treatments and interventions applied for MPN | 2 and a half months
  Type of treatments and interventions applied for MPN during COVID-19 and any change reported in therapy of MPN, particularly including:
  1. Mortality rate by discontinuation of cytoreductive drugs
  2. Mortality rate by time of exposure to cytoreductive drugs (before vs after Covid-19 pandemic)
  3. Mortality rate by cytoreductive drugs use and/or discontinuation and MPN type (MF, PV, ET, pre-PMF)
  4. Cause-specific mortality rate by cytoreductive drugs use and/or discontinuation
treatments and interventions applied for COVID-19 | 2 and a half months
  Type of treatments and interventions applied for COVID-19,
thrombotic events association to patients characteristic and treatments | 2 and a half months
  Odds Ratios (ORs) of the outcome and 95% Confidence Intervals (CIs) associated with patients' characteristics and treatments
Mortality rate occurring in the single MPN phenotypes in relation to cytoreductive treatment | 2 and a half months
  incidence of death in phenotype subgroups and by cytoreductive categories of drug
MPN progression rate | 2 and a half months
  Incidence of evolution to leukemia, myelofirbrosis and/or second cancers MPN, evaluated by cytoreductive drugs and therapy administered for COVID-19 as terms of interaction

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Barbui, Prof, Study Chair — Fondazione per la Ricerca Ospedale di Bergamo
Locations (44):
- New York-Presbyterian/Weill Cornell Medical Center, New York, New York, United States
- National Specialised Hospital for Active Treatment of Hematological Diseases, Sofia, Bulgaria
- University hospital Dubrava-School of Medicine University of Zagreb, Zagreb, Croatia
- Hopital Saint-Louis, Paris, France
- Germany (4):
  - University Hospital Halle, Department of Hematology/Oncology, Halle, Saale
  - University Medical Center RWTH, Aachen
  - University Medicine Greifswald - Hematology, Oncology, Stem Cell Transplantation and Palliative Care, Greifswald
  - University Clinic for Hematology, Oncology, Hemostaseology and Palliative Care, Johannes Wesling Medical Center, Minden
- Italy (14):
  - Ospedale San Gerardo di Monza, Monza, Monza Brianza
  - A.S.O. SS. Antonio e Biagio e C.Arrigo di Alessandria, Alessandria
  - ASST-Papa Giovanni XXIII, Bergamo
  - Policlinico S.Orsola-Malpighi, Bologna
  - ASST-Spedali Civili, Brescia
  - AOU Ospedale Careggi, Florence
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - IRCCS Policlinico San Matteo, Pavia
  - Policlinico Universitario Fondazione Agostino Gemelli, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - Ospedale Policlinico "G.B. Rossi" Borgo Roma, Verona
  - Ospedale San Bortolo, Vicenza
- Sobas Wroclaw Medical University ·, Wroclaw, Poland
- Spain (20):
  - Hospital Clínic De Barcelona, Barcelona, Barcellona
  - Hospital del Mar, Barcelona, Barcellona
  - Institut Català d' Oncologia - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - ICO L'Hospitalet - Hospital Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital General de La Palma, Breña Alta, Santa Cruz De Tenerife
  - Servicio de Hematología Hospital General Universitario de Albacete, Albacete
  - Hospital General de Elche, Alicante
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - ICO Girona Hospital Josep Trueta Servei d'hematologia, Girona
  - FEA Hematología Hospital Universitario de Móstoles, Madrid
  - Hospital 12 de octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Moncloa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario, Valencia
- Guy's and St. Thomas' NHS Foundation Trust., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Each participant can visualize its own data on eCRF after the completion patient's electronic data form.